CLINICAL TRIAL: NCT02793596
Title: Reliability of Waveform Analysis as an Adjunct to Loss of Resistance for Obstetrical Epidural Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Albert Moore, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUHC-JGH
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obstetrical patients (Experimental): Obstetrical patients requiring epidural analgesia for delivery
  Interventions: Other: Obstetrical patients

INTERVENTIONS:
Other: Obstetrical patients — Epidural waveform analysis as a confirmation of loss of Resistance

SUMMARY:
In this study, we will set out to confirm the reliability of epidural waveform analysis (EWA) as an adjunct to loss of resistance for obstetrical epidural blocks.

DETAILED DESCRIPTION:
After loss of resistance, 5 mL of normal saline will be injected through the epidural needle; the latter will then be connected to a pressure transducer (leveled with the heart) using a rigid tubing. A pressure recording of the epidural waveform will be saved for future assessment by a blinded observer.

After the recording of the waveform, the rigid tubing will be disconnected from the epidural needle. A 4 mL bolus of lidocaine 2% with epinephrine 5 µg/mL will be injected through the latter. An epidural catheter will be advanced 3-4 cm past the tip of the needle inside the epidural space. The needle will then be removed and the catheter secured to the skin in the usual fashion.

Fifteen minutes after the injection of the local anesthetic bolus, a blinded observer will apply ice to the T1-L5 dermatomes and assess the epidural block.

ELIGIBILITY:
Inclusion Criteria:

-American Society of Anesthesiologists classification 1-3

Exclusion Criteria:

* adults who are unable to give their own consent
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie transaminases ≥ 100)
* allergy to local anesthetic
* prior surgery in the lumbar spine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Success rate | 15 minutes
  Success rate evaluated with sensory block to ice

SECONDARY OUTCOMES:
Epidural waveform analysis | Immediately after epidural catheter insertion
  presence or absence of an epidural waveform measured through the epidural catheter right after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moore, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No